CLINICAL TRIAL: NCT06930105
Title: Impact of Low-Intensity Chemotherapy Combined With Short-Course Blinatumomab on Allo-HSCT in Adults With Newly Diagnosed Ph-B-ALL: A Single-Arm, Prospective, Multicenter, Phase II Study
Brief Title: Impact of Low-intensity Chemotherapy Combined With Short-course Blinatumomab on Allo-HSCT in Adults With Ph- B-ALL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xianmin Song, MD (Other)
Responsible Party: Sponsor-Investigator, Xianmin Song, MD, Director of Hematology Department, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-Blina-Ph-B ALL-2025
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Lymphoid Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blina combined low-intensity therapy (Experimental)
  Interventions: Drug: Blinatumomab plus Reduced-dose Chemotherapy

INTERVENTIONS:
Drug: Blinatumomab plus Reduced-dose Chemotherapy — Newly diagnosed Philadelphia chromosome-negative acute B-cell lymphoblastic leukemia (Ph-negative B-ALL) patients aged 18-60 years were enrolled.
  Treatment Protocol
  1. Low-intensity chemotherapy (VIP regimen)
     * V (Vincristine): 1.4 mg/m² (max 2 mg) on days 1 and 8.
     * I (Idarubicin): 8 mg/m²/day on days 1 and 8.
     * P (Prednisone): 60 mg/m²/day (max 100 mg/day) or equivalent dexamethasone dose on days 1-14.
  2. Sequential induction therapy:
     * Blinatumomab administered for 2 weeks following the VIP regimen.
  3. Consolidation therapy for morphological complete remission (CR)
     * Patients achieving CR receive two cycles of consolidation chemotherapy:
     * Cycle 1: VDCP regimen (Vincristine, Daunorubicin, Cyclophosphamide, Prednisone).
     * Cycle 2: VP + HD-MTX regimen (Vincristine, Prednisone + High-Dose Methotrexate).
  4. Allogeneic hematopoietic stem cell transplantation (allo-HSCT):
     * Patients with multiparameter flow cytometry-confirmed minimal res

SUMMARY:
This single-arm, prospective, multicenter, phase II study will enroll newly diagnosed Philadelphia chromosome-negative (Ph-) acute B-cell lymphoblastic leukemia (B-ALL) patients aged 18-60 years. Participants will receive sequential low-intensity chemotherapy followed by a two-week blinatumomab induction therapy.

Treatment Protocol

1. Low-intensity chemotherapy (VIP regimen)

   * V (Vincristine): 1.4 mg/m² (max 2 mg) on days 1 and 8.
   * I (Idarubicin): 8 mg/m²/day on days 1 and 8.
   * P (Prednisone): 60 mg/m²/day (max 100 mg/day) or equivalent dexamethasone dose on days 1-14.
2. Sequential induction therapy:

   * Blinatumomab administered for 2 weeks following the VIP regimen.
3. Consolidation therapy for morphological complete remission (CR)

   * Patients achieving CR receive two cycles of consolidation chemotherapy:
   * Cycle 1: VDCP regimen (Vincristine, Daunorubicin, Cyclophosphamide, Prednisone).
   * Cycle 2: VP + HD-MTX regimen (Vincristine, Prednisone + High-Dose Methotrexate).
4. Allogeneic hematopoietic stem cell transplantation (allo-HSCT):

   * Patients with multiparameter flow cytometry-confirmed minimal residual disease (MRD)-negative status proceed to allo-HSCT.

Patients achieving morphological complete remission (CR) will undergo two cycles of consolidation chemotherapy. Those with minimal residual disease (MRD)-negative status confirmed by multiparameter flow cytometry (MFC) or next-generation sequencing (NGS) will proceed to allogeneic hematopoietic stem cell transplantation (allo-HSCT). The primary endpoint is 18-month relapse-free survival (RFS) rate, the secondary endpoints were composite response rate (CRc: CR + CR with incomplete hematologic recovery [CRi]), MRD-negative rate (assessed by MFC/NGS),18-month overall survival (OS) post-transplant, non-relapse mortality (NRM), cumulative incidence of acute/chronic graft-versus-host disease (GVHD), cumulative relapse rate and 18-month GVHD-free/relapse-free survival (GRFS) post-transplant.

ELIGIBILITY:
Inclusion Criteria:

Patients (Age 18-60 years ) with an ECOG performance status of 0-2 and HCT-CI score <3.

2. Diagnosis: Confirmed Philadelphia chromosome-negative (Ph-) acute B-cell lymphoblastic leukemia (B-ALL) by:

* Bone marrow morphology
* Cytochemistry
* Immunophenotyping (CD19-positive by flow cytometry, ≥20% positivity on leukemic cells)
* Chromosomal analysis
* Molecular/genetic testing. 3. Planned allo-HSCT candidates must have an eligible hematopoietic stem cell donor, including:
* HLA-matched sibling donors
* Unrelated donors (9/10 or 10/10 HLA allele-matched by high-resolution typing)
* Haploidentical related donors. 4. No significant organ dysfunction:
* Liver: ALT/AST ≤3× upper limit of normal (ULN); total bilirubin ≤2× ULN.
* Kidney: BUN and serum creatinine ≤1.25× ULN.
* Cardiac:
* No acute myocardial infarction or severe arrhythmia on ECG.
* Left ventricular ejection fraction (LVEF) ≥50% on echocardiography; no significant cardiomegaly, valvular disease, or congenital heart defects.
* Pulmonary: FEV1, FVC, and DLCO ≥60% of predicted values. 5. Contraception:
* Men, women of childbearing potential (postmenopausal women must be amenorrheic for ≥12 months), and their partners must use investigator-approved effective contraception during treatment and for ≥12 months after the last study intervention.

  6. Informed consent: Patients and their legal guardians must provide written informed consent, demonstrate willingness to undergo allo-HSCT, and agree to comply with treatment protocols, follow-up schedules, and laboratory tests.

Exclusion Criteria:

1. Non-de novo patients(i.e., relapsed/refractory disease).
2. BCR-ABL1 fusion gene-positive (Ph+ ALL confirmed by molecular testing).
3. Uncontrolled active infections or viral diseases:

   * Active bacterial, viral, or fungal infections requiring treatment.
   * Hepatitis B: HBsAg-positive or HBcAb-positive with detectable HBV DNA in peripheral blood.
   * Hepatitis C: HCV antibody-positive with detectable HCV RNA.
   * Syphilis: Positive TRUST test.
   * HIV: HIV antibody-positive.
4. Major organ dysfunction or comorbidities:

   * Cardiovascular:
   * Uncontrolled hypertension, hypertensive crisis, or encephalopathy.
   * History of congestive heart failure (CHF), unstable angina, clinically significant arrhythmias (e.g., ventricular fibrillation, ventricular tachycardia).
   * Arterial thrombosis within 3 months (e.g., stroke, transient ischemic attack).
   * Symptomatic deep vein thrombosis (DVT) or pulmonary embolism (PE) within 6 months.
   * Coronary angioplasty, defibrillation, or other high-risk cardiovascular procedures.
   * Pulmonary: Severe respiratory insufficiency.
   * Gastrointestinal: Active bleeding within 3 months.
5. Uncontrolled concurrent illnesses that may compromise safety or study integrity.
6. Active or untreated central nervous system (CNS) involvement (e.g., CNS leukemia, epilepsy requiring therapy).
7. Pregnancy, lactation, or plans for pregnancy within 1 year post-infusion or during the study period.
8. Uncontrolled active infections (excluding uncomplicated UTIs or upper respiratory infections).
9. Hypersensitivity to blinatumomab or its components.
10. Inability to provide informed consent or comply with study procedures.
11. Investigator discretion: Any condition deemed to jeopardize patient safety or interfere with study objectives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
RFS | three year
  18-month relapse-free survival (RFS) rate post-allo-HSCT in newly diagnosed Ph- B-ALL patients treated with low-intensity chemotherapy followed by short-course blinatumomab induction.

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin song, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No